CLINICAL TRIAL: NCT06406647
Title: Adding Ketamine as Adjuvant in Retroclavicular Block in Upper Limb Orthopedic Surgey
Brief Title: Rectroclavicular Block in Orthopedic Surgey
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Ismail Abdelsabour, lecture of anesthesia and ICU, New Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Newvalley anesthesia
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine with bupicavaine (Active Comparator): (bupivacaine+ ketamine): 40patients received 40 ml of bupivacaine 0.25%(in total 100mg)+1mg per Kg of ketamine)
  Interventions: Other: retrocalvicular block
- bupicavacine (control group) (Active Comparator): (Bupivacaine): 40patients received40 ml of bupivacaine 0.25%(in total 100 mg)+2 ml saline.
  Interventions: Other: retrocalvicular block

INTERVENTIONS:
Other: retrocalvicular block — retrocalvicular block in upper limb orthopedic Surgey

SUMMARY:
The ultrasound-guided retroclavicular approach to the infraclavicular region (RAPTIR) brachial plexus block has gained popularity as a relatively easy-to-perform nerve block that provides reliable and dense anesthesia to the upper extremity with a single injection. The block has been well described in the anesthesia community since it was first introduced by Hebbard and Royse in 2007 . In 2017, Luftig first described the block's use in the ED setting for a variety of indications . This nerve block has classically been described to provide extensive anesthesia for procedures distal to the shoulder, such as elbow dislocations, distal radius fractures, and surgical procedures.

DETAILED DESCRIPTION:
Ultrasound-guided regional anesthesia of the infraclavicular brachial plexus offers dense anesthesia of the distal upper extremity. The Retro clavicular Approach to The Infraclavicular Region (RAPTIR) is an ultrasound-guided brachial plexus block that has only recently been described in both anesthesia and emergency literature.

Ketamine is a dissociative anesthetic used medically for induction and maintenance of anesthesia. It is also used as a treatment for depression, a pain management tool, and as a recreational drug . Ketamine is a novel compound that was derived from phencyclidine in 1962 in pursuit of a safer anesthetic with fewer hallucinogenic effects .

At anesthetic doses, ketamine induces a state of dissociative anesthesia, a trance-like state providing pain relief, sedation, and amnesia . The distinguishing features of ketamine as anesthesia are preserved breathing and airway reflexes, stimulated heart function with increased blood pressure, and moderate bronchodilation At lower, sub-anesthetic doses, ketamine is a promising agent for pain and treatment-resistant depression. As with many antidepressants, the results of a single administration of ketamine wane with time. The long-term effects of repeated use are largely unknown, and are an area of active investigation.

Liver and urinary toxicity have been reported among regular users of high doses of ketamine for recreational purposes. Ketamine is an NMDA receptor pore blocker, accounting for most of its actions, but not the antidepressant effect, the mechanism of which is a matter of research and debate.

Ketamine was first synthesized in 1962 and approved for use in the United States in 1970. It has been regularly used in veterinary medicine and was extensively used for surgical anesthesia in the Vietnam War. Along with other psychotropic drugs, it is on the World Health Organization's List of Essential Medicines. It is available as a generic medication. When used as a recreational drug, it is found both in powder and liquid form, and is often referred to as "Special K" for its hallucinogenic and dissociative effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing upper limb orthopedic surgery,

Exclusion Criteria:

* - Contraindications to regional block (coagulopathy, infection at the needle insertion site, or diaphragmatic paralysis).
* Altered conscious level.
* Pregnancy.
* Body mass index (BMI > 35).
* Patients who have difficulty understanding the study protocol.
* Patients who have any known contraindication to study medications.
* Patient refusal.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
numerical rating pain scale . | 24 hours
  0= no pain , 10 = sever pain

CONTACTS AND LOCATIONS:
Overall Officials: ahmed ismail, lecture, Principal Investigator — New Valley University
Locations (1):
- Faculty of Medicine, Asyut, Egypt